CLINICAL TRIAL: NCT02517697
Title: Nitrite Modulation of Hypertension, Platelet Activation, and Endothelial and Mitochondrial Function
Brief Title: Oral Nitrite Trial for Hypertension and Metabolic Syndrome
Acronym: ONPC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We will not initiate recruitment for this protocol due to lack of funding to support this placebo-controlled trial.
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Kara S Hughan, MD, Assistant Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO15050540
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active drug (Experimental): 14 Nitrogen (N) Sodium Nitrite 40mg three times daily (TID)
  Interventions: Drug: 14 Nitrogen (N) Sodium Nitrite
- Placebo (Placebo Comparator): placebo capsules three time daily (TID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 14 Nitrogen (N) Sodium Nitrite — oral formulation of sodium nitrite 40 mg three times daily for 12 weeks
  Other Names: sodium nitrite
  Arms: Active drug
Drug: Placebo — oral formulation of matching placebo three times daily for 12 weeks
  Arms: Placebo

SUMMARY:
The objective of the study is to investigate effects of inorganic sodium nitrite on the cardiometabolic and hormonal disturbances observed in a targeted population of overweight/obese adults with metabolic syndrome and hypertension, at risk for insulin resistance and endothelial dysfunction.

DETAILED DESCRIPTION:
Cardiovascular disease remains the leading cause of death in the United States and worldwide. Several studies have demonstrated that fruit and vegetable rich diets significantly reduced blood pressure and reduced the risk of ischemic stroke and cardiovascular disease in general, the exact mechanisms remain poorly understood. Preclinical and clinical research over the last decade has revealed the important vasoprotective effects of nitrates and nitrites with regards to reduction in blood pressure, vascular inflammation and endothelial dysfunction. More recent findings suggest that inorganic nitrate and nitrite therapy may be involved in the regulation of glucose-insulin homeostasis.

For this reason, development of an oral formulation of nitrite salt represents a rational avenue of exploration for the treatment of cardiovascular diseases, whereby nitrite would ensure rapid acting effects upon absorption. Nitrite could then be oxidized to nitrate via the enterosalivary circulation pathway. In this pathway, about 25% of circulating nitrate is concentrated in the saliva and reduced to nitrite by commensal mouth bacteria with nitrate reductase enzymes. The proposal will investigate the inorganic nitrite effects (in any form) on insulin sensitivity in a targeted population of overweight/obese adults with metabolic syndrome and hypertension, at risk for insulin resistance and endothelial dysfunction. This will be the third human trial using orally delivered nitrite (previously as aqueous solution).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Body mass index (BMI) ≥ 30 kg/m2
* Hypertension: defined as systolic blood pressure ≥130 and/or diastolic blood pressure ≥85 mm Hg
* Waist circumference: >102 cm in men, >88 cm in women

Exclusion Criteria:

* Positive urine pregnancy test or breastfeeding
* Concurrent use of medications affecting glucose metabolism (oral hypoglycemics, insulin, atypical antipsychotics)
* Recent addition or change in dosing of hormonal contraceptive medications (Oral Contraceptive Pill (OCP), Intra Uterine Device (IUD), DepoProvera shot)
* Current use of ≥3 anti-hypertensive agents regardless of blood pressure control or normotensive on a single or double agent
* Current use of phosphodiesterase-5 (PD) inhibitors or organic nitrates. We will not exclude for dietary sources of nitrate/nitrite.
* Not stable on treatments for the prior three months or not planning to remain on current dose of medications for blood pressure, contraception, etc.
* Known chronic psychiatric or medical conditions including diabetes, liver or kidney disease or obesity syndromes
* Thyroid Stimulating Hormone (TSH) >8 milli-International unit/mL
* Smoker
* Anemia (central lab hemoglobin < 11g/dL)
* Active periodontal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity (i.e. insulin stimulated glucose disposal) | baseline and 12 weeks
  obtained by hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
Change in systolic blood pressure | baseline and 12 weeks
  ambulatory blood pressure
Change in mean arterial pressure | baseline and then biweekly throughout the 12 week treatment
  ambulatory blood pressure
Change in diastolic blood pressure | baseline and 12 weeks
  ambulatory blood pressure
Change in methemoglobin level | baseline and then biweekly throughout the 12 week treatment
  by co-oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Kara S Hughan, MD, Principal Investigator — University of Pittsburgh; Mark Gladwin, MD, Study Director — University of Pittsburgh
Locations (1):
- Montefiore Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No